CLINICAL TRIAL: NCT01536704
Title: A Single Dose Bioequivalence Study of 2 Different Doses of Mini Cherry Nicotine Lozenges
Brief Title: Nicotine Lozenge Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: S6491365
Record Dates: First submitted 2011-12-15; First posted 2012-02-22 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-03

CONDITIONS: Smoking Cessation
Keywords: nicotine lozenge; nicotine; nicotine replacement therapy
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test nicotine lozenge (2 mg) (Experimental): 2 mg test nicotine lozenge to be chewed.
  Interventions: Drug: Nicotine (2 mg)
- Test nicotine lozenge (4 mg) (Experimental): 4 mg test nicotine lozenge to be chewed.
  Interventions: Drug: Nicotine (4 mg)
- Reference nicotine lozenge (2 mg) (Active Comparator): 2 mg reference nicotine lozenge to be chewed.
  Interventions: Drug: Nicotine (2 mg)
- Reference nicotine lozenge (4 mg) (Active Comparator): 4 mg reference nicotine lozenge to be chewed.
  Interventions: Drug: Nicotine (4 mg)

INTERVENTIONS:
Drug: Nicotine (2 mg) — 2 mg nicotine lozenge in two formulations
  Arms: Reference nicotine lozenge (2 mg); Test nicotine lozenge (2 mg)
Drug: Nicotine (4 mg) — 4 mg nicotine lozenge in two formulations
  Arms: Reference nicotine lozenge (4 mg); Test nicotine lozenge (4 mg)

SUMMARY:
To compare the bio equivalence of new nicotine lozenge formulation with the reference nicotine lozenge so as to deliver the same nicotine blood profile.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy smokers who usually smoked their first cigarette within 30 minutes of waking.
* Body Mass Index within the range 19-27 kilograms/meters^2

Exclusion Criteria:

* Participants who used chewing tobacco or tobacco products other than cigarettes within 21 days of screening visit

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Celerion NEBRASKA, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Out of 141 participants screened, only 50 were randomized since 91 were screen failures.
Groups:
- 2 Milligram (mg) Cherry Lozenge: Participants were instructed to move the 2mg Cherry mini nicotine lozenge from one side of the mouth to the other periodically and not to swallow or chew the lozenge.
- 2mg Mint Lozenge: Participants were instructed to move the 2mg Mint (peppermint) mini nicotine lozenge from one side of the mouth to the other periodically and not to swallow or chew the lozenge.
- 4mg Cherry Lozenge: Participants were instructed to move the 4mg Cherry mini nicotine lozenge from one side of the mouth to the other periodically and not to swallow or chew the lozenge.
- 4mg Mint Lozenge: Participants were instructed to move the 4mg Mint mini nicotine lozenge from one side of the mouth to the other periodically and not to swallow or chew the lozenge.
Period: Period 1
Arm/Group | 2 Milligram (mg) Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Started | 12 | 12 | 13 | 13
Completed | 12 | 12 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | 2 Milligram (mg) Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Started | 12 | 12 | 13 | 13
Completed | 11 | 10 | 13 | 13
Not Completed | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Period: Period 2
Arm/Group | 2 Milligram (mg) Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Started | 13 (Due to crossover design, a different set of subjects received this treatment compared to Period 1) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 1) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 1) | 13 (Due to crossover design, a different set of subjects received this treatment compared to Period 1)
Completed | 13 | 11 | 10 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | 2 Milligram (mg) Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Started | 13 | 11 | 10 | 13
Completed | 12 | 11 | 10 | 12
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | 2 Milligram (mg) Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Started | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 2) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 2) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 2) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 2)
Completed | 10 | 12 | 12 | 10
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout Period 3
Arm/Group | 2 Milligram (mg) Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Started | 10 | 12 | 12 | 10
Completed | 10 | 12 | 11 | 10
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Period 4
Arm/Group | 2 Milligram (mg) Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Started | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 3) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 3) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 3) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 3)
Completed | 12 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline measures
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 50
Age Continuous [Mean (Standard Deviation); unit: Years] | 30.3 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Time t [AUC(0-t)]
Description: AUC(0-t) was evaluated using the trapezoid rule.
Time Frame: Blood samples taken pre-dose and post-dose at 3, 5, 10, 15, 20, 30, 40, and 50 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours
Population: Analysis was done per intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: nanogram (ng).hour (hr)/millilitre (mL)
Groups:
- 2mg Cherry Lozenge: Participants were instructed to move the 2mg Cherry mini nicotine lozenge from one side of the mouth to the other periodically and not to swallow or chew the lozenge
- 4mg Mint Lozenge: Participants were instructed to move the 4mg Mint (peppermint) mini nicotine lozenge from one side of the mouth to the other periodically and not to swallow or chew the lozenge
Arm/Group | 2mg Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Number analyzed (Participants) | 47 | 45 | 45 | 47
nanogram (ng).hour (hr)/millilitre (mL) | 18.84 (7.07) | 20.71 (7.42) | 34.71 (14.48) | 33.68 (12.17)
Statistical Analysis 1: Comparison: 2mg Cherry Lozenge vs 2mg Mint Lozenge; The value was log-transformed and a linear mixed effects model was applied to this value, as the dependent variable, treatment, and period as fixed effects and participants as random effect; Test type: Non-Inferiority or Equivalence — Bio-equivalence between two dosage treatments was concluded if the 90% confidence interval for the ratio of the means for AUC (0-t) lies within the interval 0.80 to 1.25; Wilcoxon Signed Rank Test; Geometric Mean Ratio = 0.91, 90% CI 2-sided [0.88 to 0.94] — Geometric mean ratio of Cherry and Mint lozenge was determined by exponentiating least-squares means of log-transformed value
Statistical Analysis 2: Comparison: 4mg Cherry Lozenge vs 4mg Mint Lozenge; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Wilcoxon Signed Rank test; Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.98 to 1.05] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Maximum Observed Plasma Concentration [Cmaximum (Max)]
Description: Cmax was depicted from plasma concentration of nicotine.
Time Frame: as for outcome 1
Population: Analysis was done per intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 2mg Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Number analyzed (Participants) | 47 | 45 | 45 | 47
ng/mL | 5.67 (1.53) | 6.35 (1.43) | 9.37 (2.63) | 9.72 (2.70)
Statistical Analysis 1: Comparison: 2mg Cherry Lozenge vs 2mg Mint Lozenge; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Bio-equivalence between two dosage treatments was concluded if the 90% confidence interval for the ratio of the means for Cmax lies within the interval 0.80 to 1.25; Wilcoxon Signed Rank Test; Geometric Mean Ratio = 0.89, 90% CI 2-sided [0.85 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 4mg Cherry Lozenge vs 4mg Mint Lozenge; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Wilcoxon Signed Rank Test; Geometric Mean Ratio = 0.97, 90% CI 2-sided [0.93 to 1.02] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC [0-infinity (Inf)]
Description: AUC (0-inf) was evaluated using the trapezoid rule.
Time Frame: as for outcome 1
Population: Analysis was done per intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | 2mg Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Number analyzed (Participants) | 44 | 44 | 45 | 47
ng.hr/mL | 21.03 (8.05) | 22.66 (8.48) | 37.48 (16.87) | 36.08 (13.96)
Statistical Analysis 1: Comparison: 2mg Cherry Lozenge vs 2mg Mint Lozenge; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Bio-equivalence between two dosage treatments was concluded if the 90% confidence interval for the ratio of the means for AUC (0-inf) lies within the interval 0.80 to 1.25; Wilcoxon Signed Rank Test; Geometric Mean Ratio = 0.92, 90% CI [0.88 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 4mg Cherry Lozenge vs 4mg Mint Lozenge; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Wilcoxon Signed Rank Test; Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.98 to 1.06] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Reach Maximum Plasma Nicotine Concentration (Tmax)
Description: Tmax was time at which Cmax of nicotine was reached.
Time Frame: as for outcome 1
Population: Analysis was done per intention to treat (ITT) population.
Measure: Median (Full Range); unit: hr
Arm/Group | 2mg Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Number analyzed (Participants) | 47 | 45 | 45 | 47
hr | 0.83 [0.3 to 2.0] | 0.67 [0.3 to 2.0] | 0.83 [0.3 to 2.0] | 0.83 [0.3 to 2.0]
Statistical Analysis 1: Comparison: 2mg Cherry Lozenge vs 2mg Mint Lozenge; The null hypothesis considered that there is no median within-subject difference between two treatment groups; Test type: Superiority or Other; p = 0.1491, Wilcoxon Signed Rank Test; The value of Tmax was adjusted for this non-parametric analysis; Median Difference (Final Values) = 0.0006 — The median difference was calculated as Cherry minus Peppermint
Statistical Analysis 2: Comparison: 4mg Cherry Lozenge vs 4mg Mint Lozenge; The null hypothesis considered that there is no median within-subject difference between two treatment groups; Test type: Superiority or Other; p = 0.6790, Wilcoxon Signed Rank Test; The value of Tmax was adjusted for this non-parametric analysis; Mean Difference (Final Values) = 0.0005 — The median difference was calculated as Cherry minus Peppermint

5. Secondary Outcome: Apparent Elimination Half-life of Nicotine T(1/2)
Description: T(1/2) was calculated using plasma time-concentration values.
Time Frame: as for outcome 1
Population: Analysis was done per intention to treat (ITT) population.
Measure: Median (Full Range); unit: hr
Arm/Group | 2mg Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Number analyzed (Participants) | 44 | 44 | 45 | 47
hr | 3.39 [1.4 to 5.0] | 3.41 [1.4 to 6.6] | 3.19 [1.5 to 5.3] | 3.13 [1.4 to 5.3]
Statistical Analysis 1: Comparison: 2mg Cherry Lozenge vs 2mg Mint Lozenge; The null hypothesis considered that there is no median within-subject difference between two treatment groups; Test type: Superiority or Other; p = 0.5619, Wilcoxon Signed Rank Test; The value of T (1/2) was adjusted for this non-parametric analysis; Mean Difference (Final Values) = -0.0641 — The median difference was calculated as Cherry minus Peppermint
Statistical Analysis 2: Comparison: 4mg Cherry Lozenge vs 4mg Mint Lozenge; The null hypothesis considered that there is no median within-subject difference between two treatment groups; Test type: Superiority or Other; p = 0.4523, Wilcoxon Signed Rank Test; The value of T (1/2) was adjusted for this non-parametric analysis; Mean Difference (Final Values) = 0.0538 — The median difference was calculated as Cherry minus Peppermint

6. Secondary Outcome: Elimination Rate Constant for Plasma Nicotine: K (el)
Description: Kel was calculated with the help of plasma time concentration values.
Time Frame: as for outcome 1
Population: Analysis was done per intention to treat (ITT) population.
Measure: Median (Full Range); unit: 1/hr
Arm/Group | 2mg Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Number analyzed (Participants) | 44 | 44 | 45 | 47
1/hr | 0.20 [0.1 to 0.5] | 0.20 [0.1 to 0.5] | 0.22 [0.1 to 0.5] | 0.22 [0.1 to 0.5]
Statistical Analysis 1: Comparison: 2mg Cherry Lozenge vs 2mg Mint Lozenge; The null hypothesis considered that there is no median within-subject difference between two treatment groups; Test type: Superiority or Other; p = 0.5113, Wilcoxon Signed Rank Test; This non-parametric analysis was performed on the unadjusted values of parameters; Median Difference (Final Values) = 0.0025 — The median difference was calculated as Cherry minus Peppermint
Statistical Analysis 2: Comparison: 4mg Cherry Lozenge vs 4mg Mint Lozenge; The null hypothesis considered that there is no median within-subject difference between two treatment groups; Test type: Superiority or Other; p = 0.5370, Wilcoxon Signed Rank Test; This non-parametric analysis was performed on the unadjusted values of parameters; Median Difference (Final Values) = -0.0042 — The median difference was calculated as Cherry minus Peppermint

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the starting time of the investigational product, and until 5 days following last administration of the investigational product.
Arm/Group | 2mg Cherry Lozenge | 2mg Mint Lozenge | 4mg Cherry Lozenge | 4mg Mint Lozenge
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/45 | 1/47
Other Adverse Events (participants affected / at risk) | 6/47 | 9/46 | 13/45 | 15/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg Cherry Lozenge (N=47) | 2mg Mint Lozenge (N=46) | 4mg Cherry Lozenge (N=45) | 4mg Mint Lozenge (N=47)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg Cherry Lozenge (N=47) | 2mg Mint Lozenge (N=46) | 4mg Cherry Lozenge (N=45) | 4mg Mint Lozenge (N=47)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.